CLINICAL TRIAL: NCT02525380
Title: Phase4, to Assess Time to Progression (TTP) and Safety Profile of Doxorubicin-Eluting-Bead Embolization(DEBDOX) in Patients With Advanced HCC
Brief Title: Safety and Efficacy of Doxorubicin-eluting-bead Embolization in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Yoon Jun Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCbead_PVTT
Record Dates: First submitted 2015-07-29; First posted 2015-08-17 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial chemoembolization; Doxorubicin-Eluting-Bead Embolization; DC Bead TACE; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin loadeing-DC Bead(Device) (Experimental): DC Bead comprises hydrogel microspheres that are biocompatible, hydrophilic, non resorbable, precisely calibrated and capable of loading doxorubicin.
  DC Bead is produced from polyvinyl alcohol.
  Interventions: Procedure: Device(DC Bead)

INTERVENTIONS:
Procedure: Device(DC Bead) — Doxorubicin-Eluting-Bead Embolization (DEBDOX), DC Bead are a novel drug delivery embolization system

SUMMARY:
Safety and efficacy of doxorubicin-eluting-bead embolization in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) represents a first-line non-curative therapy for hepatocellular carcinoma (HCC). TACE is associated with unsatisfactory long-term outcomes. The objective response rate of TACE is only 15% to 55%, and the tumor recurrence rate is 70% at 5 years. One potential reason for this may be the increase in plasma vascular endothelial growth factor (VEGF) levels after TACE. Disturbances in the tumor microenvironment following TACE result in increased hypoxia, leading to an up-regulation in hypoxia inducible factor-1a, which in turn up-regulates VEGF and platelet-derived growth factor receptor (PDGFR) and increases tumor angiogenesis. TACE is considered for the patients with unresectable HCCs that are also ineligible for local ablative therapy. The lack of portal blood flow (because of portal vein thrombosis, portosystemic anastomoses or hepatofugal flow) had been considered as the main contraindication of TACE. However, it has been reported that TACE can be safely performed in a selected population of patients with main portal vein invasion, if they have well-preserved liver function due to collateral blood supply.

DC Beads are a novel drug delivery embolization system comprised of biocompatible, non-resorbable polyvinyl alcohol polymer hydrogel beads which can be loaded with cytotoxic drugs. The beads have a high affinity for drugs and this enables the gradual release of doxorubicin into the tumor, allowing a longer intratumoral exposure and less systemic exposure of the drug, reducing systemic toxicity. One multivariate analysis study showed that the median survival duration for the patients with portal vein invasion who were treated with DC-bead TACE (DEBDOX) were 176 days, retrospectively.

In international, multicenter, randomized phase II trial, the drug-eluting bead group showed higher rates of complete response and objective response compared with the cTACE group (27% vs. 22%, 52% vs. 44% respectively). The hypothesis of superiority was not met. However, patients with Child-Pugh B, ECOG 1, bilobar disease, and recurrent disease showed a significant increase in objective response compared to cTACE.

Here, the investigators will investigate the safety and efficacy of DC Bead TACE in patients with advanced HCC with portal vein invasion.

ELIGIBILITY:
Inclusion Criteria:[Stage C HCC according to the BarcelonaClinic of Liver Cancer]

1. Signed written informed consent.
2. Clinical or histological diagnosis of HCC based on the guidelines of the American Association for the Study of Liver Diseases.
3. At least one typical enhanced lesion that is bi-dimensionally measurable by multiphasic spiral CT scan or dynamic contrast-enhanced MRI.
4. Tumor conditions confirmed by abdominal imaging (contrast enhanced CT ± MRI) performed within 1 month prior to the enrollment:
5. Age of at least 18 years and less than 80 years.
6. ECOG Performance Status of 0 or 1.
7. Child-Pugh class A or B (Child-Pugh score ≤ 7).
8. Life expectancy of at least 16 weeks.
9. Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements (no transfusion, no restoration), conducted within 14 days prior to screening:

   * Hemoglobin ≥ 8.0 g/dL
   * Absolute neutrophil count ≥ 1,000/mm3
   * Platelet count ≥ 50,000/μL
   * Total bilirubin <2.5 mg/dL
   * Serum albumin ≥2.8 g/dL
   * ALT and AST < 5 × upper limit of normal
   * PT-INR ≤ 2.3 or Prothrombin Time-sec ≤ 6 sec
   * Serum creatinine ≤ 1.7 mg/dL

Exclusion Criteria:

1. A history of receiving any systemic therapy of the molecularly targeted agents, immunotherapy or cytotoxic chemotherapy for the treatment of HCC
2. Invasion of inferior vena cava (Vv3), or invasion of first order branch of the biliary duct (B3)
3. History or presence of hepatic encephalopathy
4. Ascites, moderate, large or intractable
5. Active clinically serious infections (> grade 2, NCI-CTC version 4.0), including spontaneous bacterial peritonitis.
6. Untreated active chronic hepatitis B
7. Esophageal or gastric varices≥ F2 (grade 2) with red color sign positive without prophylaxis (non-selective beta-blocker or endoscopic variceal ligation) or history of variceal bleeding without endoscopic variceal ligation/ injection sclerosis
8. Active ulcer of stomach or duodenum: untreated or presence of visible vessel
9. Any major surgery within 4 weeks, or any minor surgery within 2 weeks prior to signing the informed consent form
10. Candidate for liver transplant and a history of liver transplantation
11. History of cardiac disease: congestive heart failure greater than NYHA class 2; active coronary artery disease; cardiac arrhythmias requiring anti-arrhythmic therapy or uncontrolled hypertension and diabetes mellitus
12. History of AIDS/HIV infection.
13. Seizure disorder requiring medication.
14. History of organ allograft.
15. Evidence or history of bleeding diathesis, or thromboembolic events requiring treatment
16. Current renal dialysis.
17. Previous or concurrent cancer that has a primary site or histology distinct from HCC, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis, and T1] or any cancer curatively treated less than 3 years prior to enrollment.
18. History of alcohol abuse (male > 210g/week, female >140g/week)
19. Any contraindication for chemoembolization except major branch of portal vein invasion
20. Any contraindication for doxorubicin administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
The rate of Time to progression of hepatocellular carcinoma 30 patients. | up to at least 3 years
  The rate of Time to progression of doxorubicin eluting bead embolization in patients with advanced hepatocellular carcinoma.After the treatment period, patients will undergo follow up for safety within 30 days (+7 days) of final DEBDOX, and will undergo follow up for survival every 84 days (±14 days) (84 days is the day counted from the DEBDOX TACE) for at least 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea